CLINICAL TRIAL: NCT00519753
Title: Safety and Efficacy of Switching to the Travoprost/Timolol Maleate Fixed Combination (DUOTRAV®) From Prior Mono or Two-Drug Therapy in Germany
Brief Title: Success of Transitioning Uncontrolled Glaucoma Patients From Prior Mono or Adjunctive Therapy to DuoTrav
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMS-06-12
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2010-01

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Travoprost; Timolol; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DuoTrav (Experimental): One drop in study eye(s) once daily in the evening (at 8:00 PM) for 12 weeks
  Interventions: Drug: Travoprost 0.004%/timolol maleate 0.5% fixed combination ophthalmic solution (DuoTrav)

INTERVENTIONS:
Drug: Travoprost 0.004%/timolol maleate 0.5% fixed combination ophthalmic solution (DuoTrav) — One drop in study eye(s) once daily in the evening (at 8:00 PM) for 12 weeks
  Other Names: DUOTRAV®

SUMMARY:
The purpose of this study is to assess the safety and efficacy of transitioning uncontrolled glaucoma patients to DuoTrav from other mono or adjunctive therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults with primary open-angle glaucoma, ocular hypertension or pigment dispersion glaucoma.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Age related.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in intraocular pressure at 12 weeks from travoprost prior therapy (baseline) | Baseline and 12 weeks

SECONDARY OUTCOMES:
Change in intraocular pressure at 12 weeks from other prior therapies (baseline) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Jasek, Study Director — Alcon Research
Locations (1):
- Mainz, Mainz, Germany

REFERENCES:
- [Result] Pfeiffer N, Scherzer ML, Maier H, Schoelzel S, Jasek MC, Stewart JA, Stewart WC. Safety and efficacy of changing to the travoprost/timolol maleate fixed combination (DuoTrav) from prior mono- or adjunctive therapy. Clin Ophthalmol. 2010 May 14;4:459-66. doi: 10.2147/opth.s10694. PMID 20505839